CLINICAL TRIAL: NCT04616183
Title: Open-Label Phase 1b/2 Study of Cetuximab Administered in Combination With LY3214996 (ERK 1/2 Inhibitor) or Cetuximab in Combination With LY3214996 and Abemaciclib in Patients With Metastatic, Anti-EGFR-Refractory Colorectal Cancer
Brief Title: LY3214996 and Cetuximab Alone or in Combination With Abemaciclib for the Treatment of Unresectable or Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1016; NCI-2020-06350 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1016 (Other: M D Anderson Cancer Center); R01CA187238 (NIH)
Record Dates: First submitted 2020-08-31; First posted 2020-11-04 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colon Adenocarcinoma; Metastatic Colorectal Carcinoma; Metastatic Rectal Adenocarcinoma; Recurrent Colorectal Carcinoma; Stage III Colon Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Colon Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIA Rectal Cancer AJCC v8; Stage IIIB Colon Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Colon Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IIIC Rectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8; Stage IVA Colon Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8; Unresectable Colon Adenocarcinoma; Unresectable Colorectal Carcinoma; Unresectable Rectal Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Rectal Neoplasms | interventions — abemaciclib; Cetuximab; LY3214996

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (ERK1/2 inhibitor LY3214996, cetuximab) (Experimental): Patients receive ERK1/2 inhibitor LY3214996 PO QD on days 1-28 and cetuximab IV over 1-2 hours on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Drug: ERK1/2 Inhibitor LY3214996
- Arm B (ERK1/2 inhibitor LY3214996, cetuximab, abemaciclib) (Experimental): Patients receive ERK1/2 inhibitor LY3214996 and cetuximab as in Arm A. Patients also receive abemaciclib PO BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib; Biological: Cetuximab; Drug: ERK1/2 Inhibitor LY3214996

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY-2835219; LY2835219; Verzenio
  Arms: Arm B (ERK1/2 inhibitor LY3214996, cetuximab, abemaciclib)
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Drug: ERK1/2 Inhibitor LY3214996 — Given PO
  Other Names: LY 3214996; LY3214996

SUMMARY:
This phase Ib/II trial investigates the side effects and best dose of LY3214996 when given together with cetuximab alone or in combination with abemaciclib and to see how well they work in treating patients with colorectal cancer that cannot be removed by surgery (unresectable) and/or has spread to other places in the body (metastatic). Cetuximab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. LY3214996 and abemaciclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving LY3214996 and cetuximab alone or in combination with abemaciclib may help treat patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of ERK1/2 inhibitor LY3214996 (LY3214996) administered in combination with cetuximab. (Phase 1b) II. Determine the MTD and RP2D of LY3214996 administered in combination with cetuximab plus abemaciclib. (Phase 1b) III. Assess the preliminary antitumor activity of the treatment combinations based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. (Phase 2)

SECONDARY OBJECTIVES:

I. Assess the preliminary antitumor activity of the treatment combinations based on RECIST v.1.1. (Phase 1b) II. Characterize the safety profile of the treatment combinations (DLTs). III. Evaluate for pERK and Ki67 inhibition.

EXPLORATORY OBJECTIVES:

I. Assess blood- and tissue-based predictive biomarkers of activity and immune effects upon treatment with cetuximab, LY3214996, and abemaciclib.

II. Demonstrate feasibility of establishing patient-derived xenograft (PDX) models in matched patients with cetuximab-refractory metastatic colorectal cancer (mCRC) to evaluate for biomarkers of response and mechanisms of resistance.

III. Explore mechanisms of resistance to cetuximab plus LY3214996 and cetuximab, LY3214996, plus abemaciclib.

OUTLINE: This is a phase Ib, dose-escalation study of ERK1/2 inhibitor LY3214996 followed by a phase II study. Patients are assigned to 1 of 2 arms.

ARM A: Patients receive ERK1/2 inhibitor LY3214996 orally (PO) once daily (QD) on days 1-28 and cetuximab intravenously (IV) over 1-2 hours on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive ERK1/2 inhibitor LY3214996 and cetuximab as in Arm A. Patients also receive abemaciclib PO twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed Informed Consent prior to any screening procedures being performed. The informed consent process will be conducted in accordance with MD Anderson Office of Clinical Research SOP 04 and as indicated in Appendix 2.
* Age ≥18 years at the time of informed consent.
* Histologically (or cytologically) confirmed diagnosis of adenocarcinoma of the colon or rectum, with clinical confirmation of unresectable and/or metastatic disease that is measureable according to RECIST1.1 criteria.
* Baseline tissue-based KRAS, NRAS, EGFR, BRAF wild-type tumor. If MEK1 was tested, must be wild-type tumor
* Prior treatment with at least one systemic chemotherapy regimen for mCRC, or recurrence/progression with development of unresectable or metastatic disease within 6 months of adjuvant chemotherapy for resected colorectal cancer.
* Participants who received chemotherapy must have recovered (Common Terminology Criteria for Adverse Events [CTCAE] Grade .1) from the acute effects of chemotherapy except for residual alopecia or Grade 2 peripheral neuropathy prior to randomization. A washout period of at least 21 days is required between last chemotherapy dose and randomization (provided the participant did not receive radiotherapy).
* Participants who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization
* Left-sided primary tumor
* Prior treatment with, and progression on, anti-EGFR therapy (cetuximab or panitumumab).
* ECOG performance status ≤ 1.
* Adequate bone marrow, organ function and laboratory parameters:
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L,
* Hemoglobin (Hgb) ≥ 9 g/dL with or without transfusions,
* Platelets (PLT) ≤ 100 x 109/L without transfusions,
* AST and/or ALT ≤ 2.5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x ULN and < 2 mg/dL Note: Participants who have a total bilirubin level > 1.5 x ULN will be allowed if their indirect bilirubin level is ≤ 1.5 x ULN
* Serum Creatinine ≤ 1.5 x ULN, or calculated creatinine clearance (determined as per Cockcroft-Gault) ≥ 50mL/min at screening.
* QTc interval ≤ 480 ms (preferably the mean from triplicate ECGs);
* Able to take oral medications.
* Female participants are either postmenopausal for at least 1 year, are surgically sterile for at least 6 weeks, or must agree to take appropriate precautions to avoid pregnancy from screening through follow-up if of childbearing potential.

Note: Permitted contraception methods include: male condom with spermicide, female condom with spermicide, diaphragm with spermicide, cervical sponge, or cervical cap with spermicide. Also see the definition of highly effective method of contraception in Appendix 1. These should be communicated to the participants and their understanding confirmed. For all females, the pregnancy test result must be negative within 24 hours of starting treatment on study and within 24 hours prior to each cycle. Males must agree to take appropriate precautions to avoid fathering a child from screening through 100 days following the end of therapy.

Exclusion Criteria:

* History of a Grade 3 or 4 allergic reaction or intolerability attributed to cetuximab.
* Right-sided or transverse colonic primary tumor.
* Baseline tissue-based KRAS, NRAS, EGFR, BRAF and MEK1 mutated tumor
* Active infection requiring concurrent antibiotic use.
* Currently using concomitant medications that are strong inhibitors or inducers of CYP3A4.
* Previously completed or withdrawn from this study or any other study investigating an ERK1/2 inhibitor.
* Any known symptomatic brain metastasis. Note: Participants previously treated or untreated for this condition who are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed. Known brain metastases must be stable for ≥ 4 weeks, with imaging (e.g., magnetic resonance imaging [MRI] or computed tomography [CT]) demonstrating no current evidence of progressive brain metastases at screening.
* Known leptomeningeal disease
* Previous or concurrent malignancy within 3 years of study entry, with the following exceptions: adequately treated basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, or other noninvasive or indolent malignancy; other solid tumors treated curatively without evidence of recurrence for at least 3 years prior to study entry.
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) <6 months prior to screening,
  * Symptomatic chronic heart failure (i.e. Grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality <6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia;
  * The participant has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Uncontrolled hypertension defined as persistent elevation of systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mm Hg, despite current therapy;
* The participant has active systemic bacterial infection (requiring intravenous (IV) antibiotics at time of initiating study treatment,) fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C (for example, hepatitis B surface antigen positive.) Screening is not required for enrollment.; Known history of acute or chronic pancreatitis (history of acute pancreatitis with no recurrent events in the prior 24 months are permitted)
* Impaired gastrointestinal function or disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption).
* Any other condition that would, in the Investigator's judgment, contraindicate the participants participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* For participants receiving abemaciclib: The participant has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Major surgery ≤ 6 weeks prior to starting study drug or failure to recover from side effects of such procedure at the discretion of the treating investigator.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Best overall response (complete response [CR] + partial response [PR]) | From the start of the treatment until disease progression, assessed up to 1 year
  Response rate will be calculated based on the number of patients in the evaluable population experiencing a radiographic response according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria (either CR or PR) relative to the total number of patients in the efficacy evaluable population. A 95% confidence interval will be estimated around this population.

SECONDARY OUTCOMES:
Overall survival | From enrollment until death, assessed up to 1 year
  The Kaplan-Meier method will be used to estimate both the survival curves and the median survival time. The 95% confidence intervals for median survival times will also be calculated.
Progression-free survival (PFS) | From enrollment until death or disease progression as defined by RECIST version 1.1 criteria for the evaluable population, assessed up to 1 year
  The Kaplan-Meier method will be used to estimate the proportion of subjects without progression or death overtime and the median PFS. The 95% confidence intervals for median PFS will also be displayed.
Incidence of adverse events | Up to 30 days
  Will be tabulated for adverse events according to Common Terminology Criteria for Adverse Events version 5.0 across all grades.

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Parseghian, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT04616183/ICF_000.pdf